CLINICAL TRIAL: NCT01593722
Title: Comparison Between the Post-Treatment Reactions After Single-dose Ivermectin or DEC in Subjects With Loa Loa Infection
Brief Title: Post-treatment Effects of Ivermectin (IVM) or Diethylcarbamazine (DEC) in Loiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 999912117; 12-I-N117 (Other: NIAID IRB)
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Loiasis
Keywords: Loa loa; Immune Response; Therapy
MeSH Terms: conditions — Loiasis | interventions — Diethylcarbamazine; Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diethylcarbamazine (Active Comparator): diethylcarbamazine 8 mg/kg single oral dose
  Interventions: Drug: Diethylcarbamazine
- ivermectin (Active Comparator): ivermectin 200 mcg/kg single oral dose
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Diethylcarbamazine — single dose
  Other Names: Hetrazan, Banocide
  Arms: diethylcarbamazine
Drug: Ivermectin — single dose
  Other Names: Mectizan, Stromectol
  Arms: ivermectin

SUMMARY:
Background:

* Loa loa is a small worm that infects people in West and Central Africa. It is spread by the bite of a fly. Adult worms live under the skin and can cause swelling in the arms, legs, and face. Some people have more serious infections in the heart, kidneys, or brain. Most people with Loa loa infection have no symptoms at all. The standard treatment for Loa loa infection is a medicine called diethylcarbamazine (DEC). Some people have bad reactions to DEC, including itching, muscle pains, and in severe cases coma and death.
* Another drug, ivermectin, is used in mass drug treatment programs to prevent the spread of worm infections that cause blindness and massive swelling (elephantiasis). However, people who also have Loa loa have had serious bad reactions to ivermectin. Researchers want to study both DEC and ivermectin to find out why these reactions occur. If they can be prevented, mass drug treatment programs will be able to be used in areas in Africa where Loa loa exists.

Objectives:

- To study the side effects of DEC and ivermectin treatment for Loa loa infection.

Eligibility:

- Individuals who live in 4 villages in Cameroon where Loa loa infection is known to exist, who are between 20 and 60 years of age, not pregnant or breastfeeding and have a low level of Loa loa parasites in the blood, but are otherwise healthy.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected to check for Loa loa infection. Participants will also have an eye exam and provide skin samples to check for other worm infections that may interfere with the study treatment.
* Participants will be admitted to the hospital for 4 days (during and after the treatment). They will receive a single dose of either DEC or ivermectin.
* After treatment, regular blood samples will be collected. Participants will be asked questions about how they feel after treatment. Physical exams will be performed. If side effects develop, participants will be treated at the hospital.
* After leaving the hospital, participants will have followup visits. These visits will happen on days 5, 7, 9, and 14 after receiving the study medicine. They will involve a short physical exam and collection of blood samples.
* At the end of the study, participants will be offered a full 21-day DEC treatment to cure the Loa loa infection.

DETAILED DESCRIPTION:
Ivermectin is currently used for mass drug distribution for the control of onchocerciasis and elimination of lymphatic filariasis in Africa. Due to the occurrence of severe neurologic adverse events in individuals with concomitant Loa loa infection and high levels of circulating microfilariae, drug distribution has been halted in many areas in Cameroon, Democratic Republic of Congo and other Loa-endemic countries. Diethylcarbamazine citrate (DEC) is the treatment of choice for Loa loa infection in the United States and other non-endemic countries, but can also be associated with the development of severe adverse reactions, including fatal encephalopathy, that are correlated with the number of circulating microfilariae in the blood. The cause of these reactions is unknown, and it is not known if post-treatment reactions to DEC and ivermectin both have the same underlying mechanism. Post-treatment reactions to both medications are accompanied by a dramatic interleukin-5 (IL-5)-dependent increase in eosinophilia and evidence of eosinophil activation. Preliminary data suggests that, unlike post-treatment responses in Wolbachia-containing filariae, inflammatory mediators commonly seen in bacterial infections and malaria, including tumor necrosis factor (TNF)-alpha and IL-1-beta, are not increased post-treatment with DEC. The aim of this study is to characterize the immunologic mechanisms of ivermectin and DEC posttreatment reactions so that it can be established whether or not these posttreatment reactions have the same underlying mechanism. An understanding of the pathophysiology of these post-treatment reactions is necessary in order to develop strategies to prevent these reactions in the future. We plan to randomize 20 subjects with low- to- moderate numbers of circulating Loa loa microfilariae to receive a single oral dose of either ivermectin (200 mcg/kg) or DEC (8 mg/kg) in an inpatient setting in Cameroon. Signs and symptoms, blood microfilarial levels, complete blood counts, intracellular and serum cytokine levels and markers of eosinophil activation will be assessed at baseline, 4 and 8 hours, and 1, 2, 3, 5, 7, and 9 and 14 days post-treatment and compared between the two treatment groups. Subjects who received ivermectin will be treated with single dose DEC (8 mg/kg) on day 14. All subjects will then be followed at 6 and 12 months post-hospitalization to determine whether they have experienced Loa-specific symptoms (eyeworm or Calabar swellings). Mf count and complete blood count (CBC) with differential will be obtained at each follow-up visit. Subjects with Loa-specific symptoms or mf counts > 100 mf/mL at the 6 month time point will be offered a full treatment course. If > 50% of subjects meet criteria for full DEC treatment at the 6, month time point, all subjects will be treated and the study will enter a follow-up phase with a visit at 12 months (6 months after the full treatment course ).

ELIGIBILITY:
* INCLUSION CRITERIA (SCREENING):

A subject will be eligible for participation in the screening portion of this protocol if all of the following criteria apply:

1. male or non-pregnant and not breastfeeding female subjects,
2. age 20-60 years (per participant self-report)
3. resident of Akonolinga
4. Loa microfilaremia from 20 to 5000 mf/mL from the prior screening in the village or did not participate in the prior screening
5. consent to a blood draw to screen for infection with Loa loa
6. must be willing to have blood samples stored

EXCLUSION CRITERIA (SCREENING):

A subject will not be eligible for participation in the screening portion of this study if any of the following conditions apply:

1. Known to be pregnant (by history) or breastfeeding
2. Chronic medical conditions, including but not limited to diabetes, renal or hepatic insufficiency, immunodeficiency, psychiatric disorder, seizure, that in the investigators judgments are deemed to be clinically significant
3. History of hypersensitivity reaction to DEC or IVM

INCLUSION CRITERIA (INTERVENTIONAL STUDY):

A subject will be eligible for participation in the interventional portion of the study only if all of the following additional inclusion criteria apply:

1. Loa loa microfilaremia between 20 and 2,000 mf/mL blood drawn between 11:30 am and 2:30 pm measured within 30 days prior to the baseline visit
2. The subject agrees to storage of samples for study

EXCLUSION CRITERIA (INTERVENTIONAL STUDY):

A subject will not be eligible to participate in the interventional portion of the study if any of the following conditions are fulfilled at the time of enrollment:

1. Pregnancy (by serum or urine beta-HCG) or breastfeeding
2. Chronic kidney or liver disease
3. Hgb < 10 gm/dL
4. Filarial infection other than Loa loa or M. perstans (O. volvulus, or W. bancrofti)
5. Use of DEC or IVM within the past 6 months
6. Use of immunosuppressive therapies, including steroids, within the past month
7. Any condition that in the investigator s opinion places the subject at undue risk by participating in the study

EXCLUSION OF CHILDREN AND PREGNANT WOMEN:

Pregnant women and children (the age of consent in Cameroon is 20 years of age) will be excluded from this study since it involves administration of medications contraindicated in pregnancy and more than minimal risk with no prospect of direct benefit, respectively.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Filariasis and other Tropical Diseases Research Center, Yaoundé, Cameroon

REFERENCES:
- [Background] Klion AD, Massougbodji A, Sadeler BC, Ottesen EA, Nutman TB. Loiasis in endemic and nonendemic populations: immunologically mediated differences in clinical presentation. J Infect Dis. 1991 Jun;163(6):1318-25. doi: 10.1093/infdis/163.6.1318. PMID 2037798
- [Background] Boussinesq M. Loiasis. Ann Trop Med Parasitol. 2006 Dec;100(8):715-31. doi: 10.1179/136485906X112194. PMID 17227650
- [Background] Winkler S, Paiha S, Winkler H, Graninger W, Marberger M, Steiner GE. Microfilarial clearance in loiasis involves elevation of Th1 and Th2 products and emergence of a specific pattern of T-cell populations. Parasite Immunol. 1996 Sep;18(9):479-82. doi: 10.1111/j.1365-3024.1996.tb01032.x. PMID 9226684
- [Derived] Herrick JA, Legrand F, Gounoue R, Nchinda G, Montavon C, Bopda J, Tchana SM, Ondigui BE, Nguluwe K, Fay MP, Makiya M, Metenou S, Nutman TB, Kamgno J, Klion AD. Posttreatment Reactions After Single-Dose Diethylcarbamazine or Ivermectin in Subjects With Loa loa Infection. Clin Infect Dis. 2017 Apr 15;64(8):1017-1025. doi: 10.1093/cid/cix016. PMID 28329346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the155 subjects recruited, 92 were eligible for screening and signed consent. Thirty had loiasis, of which 16 were excluded because their microfilarial counts were >5000 mf/mL. One subject was excluded because of age and one declined to participate. The remaining 12 patients were enrolled in the treatment arm of the study.
Groups:
- Single Dose DEC: diethylcarbamazine 8 mg/kg single oral dose
  Diethylcarbamazine: single dose
- Single Dose IVM: ivermectin 200 mcg/kg single oral dose
  Ivermectin: single dose
Period: Overall Study
Arm/Group | Single Dose DEC | Single Dose IVM
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose DEC | SIngle Dose IVM | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 44.5 [20 to 60] | 38.5 [25 to 53] | 44.5 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Cameroon | 6 | 6 | 12
Absolute eosinophil count [Geometric Mean (Full Range); unit: cells x 10^9/L] | 3.27 [2.3 to 5.76] | 1.76 [1.05 to 2.35] | 2.40 [1.05 to 5.76]
Loa microfilarial count [Geometric Mean (Full Range); unit: mf/ml] | 1074 [200 to 20380] | 355 [60 to 2300] | 618 [60 to 20380]

OUTCOME MEASURES:

1. Primary Outcome: The Peak % of Baseline Eosinophil Count Measured During the First 7 Days Post-treatment.
Time Frame: 7 days
Measure: Geometric Mean (Full Range); unit: percentage of baseline
Arm/Group | Diethylcarbamazine | Ivermectin
Number analyzed (Participants) | 6 | 6
percentage of baseline | 196 [112 to 224] | 165 [124 to 257]
Statistical Analysis 1: Comparison: Diethylcarbamazine vs Ivermectin; Test type: Superiority or Other; p = 0.68, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: The Frequency of Adverse Events
Description: Symptoms, signs and laboratory abnormalities occurring in the 7 days post-treatment
Time Frame: 7 days
Measure: Number; unit: events
Arm/Group | Diethylcarbamazine | Ivermectin
Number analyzed (Participants) | 6 | 6
events | 115 | 103

3. Secondary Outcome: Eosinophil Activation
Description: Levels of surface marker expression on eosinophils
Time Frame: 3 days
Measure: Geometric Mean (Full Range); unit: % cells expressing CD69
Arm/Group | Single Dose DEC | Single Dose IVM
Number analyzed (Participants) | 6 | 6
% cells expressing CD69
  %CD69 expression on eosinophils at peak | 21.5 [6.1 to 79.7] | 21.5 [8.4 to 94]
  %CD69 expression on eosinophils at baseline | 1.7 [0.1 to 4.2] | 1.5 [0.1 to 4.6]

4. Secondary Outcome: Proportion of Subjects Who Clear Microfilaremia
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Diethylcarbamazine | Ivermectin
Number analyzed (Participants) | 6 | 6
participants | 3 | 0

5. Other Pre Specified Outcome: Treatment Efficacy
Description: Proportion of subjects without signs of infection
Time Frame: 6 months
Population: Microfilarial count and symptoms
Measure: Number; unit: participants
Arm/Group | Diethylcarbamazine | Ivermectin
Number analyzed (Participants) | 6 | 6
participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Diethylcarbamazine | Ivermectin
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diethylcarbamazine (N=6) | Ivermectin (N=6)
Calabar swelling (Skin and subcutaneous tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 4 | 4
Eyeworm (Infections and infestations) | 1 | 2
Blurry vision (Eye disorders) | 3 | 1
Paresthesia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 4 | 2
Myalgia/arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Diarrhea (Gastrointestinal disorders) | 1 | 3
Nausea/vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Palpitations (Cardiac disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Chest pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Hives (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4
Fatigue (General disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No